CLINICAL TRIAL: NCT06226480
Title: Development and Validation of a Prediction Model for Postoperative Delirium in Elderly Patients After Thoracic Surgery
Brief Title: Machine Learning Algorithm for Predicting Postoperative Delirium in Elderly Patients After Thoracic Surgery
Acronym: POD
Status: Completed | Type: Observational
Sponsor: Affiliated Hospital of Nantong University (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-K002-01; YJXYY202204-YSC07 (Other Grant/Funding Number: Jiangsu Provincial Research Hospital); QNZ2023004 (Other Grant/Funding Number: Nantong municipal health commission)
Record Dates: First submitted 2024-01-18; First posted 2024-01-26 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-01

CONDITIONS: Postoperative Delirium
Keywords: postoperative delirium
MeSH Terms: conditions — Emergence Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Postoperative delirium (POD) is a common and severe complication in patients undergoing major surgery, especially in the elderly. POD has been proven to be associated with increased morbidity and mortality, institutionalization, and high healthcare costs. This retrospective cohort study aimed to use machine learning methods to develop clinically meaningful models to support clinical decision making.

DETAILED DESCRIPTION:
The primary outcome was the incidence of POD within 3 days postoperatively. The patients will be randomly split into two datasets with split ratios of 80% and 20%.

Subsequently, 80% of the patients will be used for training, and 20% of the patients will be used for testing. Multiple machine learning algorithms will be used to develop POD risk prediction models. The discrimination ability of the prediction models will be assessed by calculating the area under the receiver operating characteristic curve (AUC). The calibration of the model will be evaluated using the Hosmer-Lemeshow goodness of fit test. Decision curve analysis (DCA) will be used to evaluate the net benefits for each threshold probability. The best model will be selected by comparing the performance between the models. Then the SHapley Additive exPlanations (SHAP) will be used to explain the best one.

ELIGIBILITY:
Inclusion Criteria:

* aged ≥ 65 years
* elective segmentectomy, lobectomy, or esophagectomy surgeries
* general anesthesia

Exclusion Criteria:

* surgery length less than 1 hour
* preoperative cognitive dysfunction
* admission to the intensive care unit
* second operation within 24 hours
* missing data for any variables

Min Age: 65 Years | Sex: All
Age Groups: Older Adult
Study Population: Elderly patients undergoing thoracic surgeries.
Sampling Method: Non-Probability Sample
Enrollment: 3967 (Actual)
Dates: Start 2024-02-25 (Actual); Primary Completion 2024-07-20 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Number of participants with postoperative delirium | The first three postoperative days
  The following descriptive words and the derivatives were searched from the medical records: "delirium", "agitation", "hallucinations", "combative behavior", "inattention", "confusion", "mental status change", "disorientation", "drowsy". Medical records with the presence of these keywords were reviewed by an independent researcher, and medical records presented the aforementioned symptoms preoperatively were excluded. Postoperative delirium was diagnosed according to the Diagnostic and Statistical Manual of Mental Disorders, fourth edition (DSM-IV) criteria.

CONTACTS AND LOCATIONS:
Locations (1):
- Affiliated Hospital of Nantong University, Nantong, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No
Only IPD used in the results publication will be shared upon reasonable request